CLINICAL TRIAL: NCT02988583
Title: Emulsification of Different Viscosity Silicone Oil After Complicated Retinal Detachment Surgery: A Randomized Double-masked Clinical Trial
Brief Title: Emulsification of Different Viscosity Silicone Oil After Complicated Retinal Detachment Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE591018
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Retinal Detachment Rhegmatogenous
Keywords: silicone oil; emulsification; retinal detachment surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low viscosity silicone oil (Experimental): Retinal detachment surgery using low viscosity silicone oil
  Interventions: Device: Surgery using low viscosity silicone oil
- high viscosity silicone oil (Active Comparator): Retinal detachment surgery using high viscosity silicone oil
  Interventions: Device: Surgery using high viscosity silicone oil

INTERVENTIONS:
Device: Surgery using low viscosity silicone oil — Pars plans vitrectomy using low viscosity silicone oil
  Arms: low viscosity silicone oil
Device: Surgery using high viscosity silicone oil — Pars plans vitrectomy using high viscosity silicone oil
  Arms: high viscosity silicone oil

SUMMARY:
Silicone oil has been used as a surgical tool in complicated retinal detachment surgery. There are some complications occurring in pars plana vitrectomy with silicone oil tamponade. Silicone oil emulsification is one of the complication that may result in severe sequels that are difficult to treat. It is believed that low viscosity silicone oil has more risk to develop emulsification than high viscosity silicone oil. Up to now, however, there is no conclusive guideline that which types of silicone oil is suitable for these complicated retinal detachment surgeries and what is the appropriate time to remove the oil. This prospective study aims to study the silicone oil emulsification comparing between low viscosity and high viscosity silicone oil after complicated retinal detachment surgery.

DETAILED DESCRIPTION:
Silicone oil has been used as a surgical tool in retinal detachment surgery since 1962. The National Eye Institute Silicone Study demonstrated the superiority of silicone oil compared with sulfur hexafluoride, and its comparability with perfluoropropane, for the treatment of complicated retinal detachment associated with advanced proliferative vitreoretinopathy. There are some complications occurring in pars plana vitrectomy with silicone oil tamponade. These complications may occur during surgery and after the surgery. Silicone oil emulsification is one of the complication that may result in severe sequels including band-shaped keratopathy, complicated glaucoma and retinopathy that are difficult to treat. The commonly used silicone oil includes low viscosity and high viscosity type. It is believed that low viscosity silicone oil has more risk to develop emulsification than high viscosity silicone oil. Up to now, however, there is no conclusive guideline that which types of silicone oil is suitable for these complicated retinal detachment surgeries and what is the appropriate time to remove the oil. Retrospective medical review of these patients using 1000-vs 5000-centistoke silicone oil demonstrated that anatomic and visual acuity outcomes, as well as complication rates including emulsification, were similar in both groups. To the best of authors' knowledge, there has been no prospective study on this subject. This study aims to study the silicone oil emulsification comparing between low viscosity and high viscosity silicone oil after complicated retinal detachment surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of complicated retinal detachment who underwent pars plana vitrectomy with intravitreal silicone oil tamponade
* Age ≥ 18 years
* Sign informed consent form

Exclusion Criteria:

* Inflammatory eye diseases i.e. uveitis
* Corneal scar
* History of scleral buckling procedure
* History of using surfactant drugs
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Emulsification rate | 12 months
  Proportion of patients developing silicone oil emulsification in each arm/group.

SECONDARY OUTCOMES:
Retina reattachment rate | 12 months
  Proportion of patients having retinal reattachment after surgery in each arm/group.
visual improvement | 12 months
  Proportion of patients having visual improvement after surgery in each arm/group

CONTACTS AND LOCATIONS:
Locations (1):
- Srinagarind Hospital, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387
- [Derived] Ratanapakorn T, Thongmee W, Meethongkam K, Sinawat S, Sanguansak T, Bhoomibunchoo C, Laovirojjanakul W, Yospaiboon Y. Emulsification of Different Viscosity Silicone Oil in Complicated Retinal Detachment Surgery: A Randomized Double-Blinded Clinical Trial. Clin Ophthalmol. 2020 Feb 7;14:359-367. doi: 10.2147/OPTH.S242804. eCollection 2020. PMID 32103882